CLINICAL TRIAL: NCT05614700
Title: Reirradiation Options for Previously Irradiated Prostate Cancer (RO-PIP): Feasibility Randomised Clinical Trial Investigating Toxicity Outcomes Following Reirradiation With Ultra-hypofractionated External Beam Radiotherapy vs. High Dose Rate Brachytherapy
Brief Title: Prostate Reirradiation Toxicity Outcomes Feasibility Study
Acronym: RO-PIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Ann Henry, Associate Professor in Clinical Oncology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/YH/0305
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries | interventions — Brachytherapy

STUDY DESIGN:
Intervention Model Description: Randomised Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose-rate brachytherapy (Active Comparator): Two HDR-BT treatment schedules, either a single fraction 19Gy treatment or 27Gy in 2 fractions approximately 2 weeks apart will be used to be decided by treating centre.
  Interventions: Radiation: Brachytherapy
- Ultra-hypofractionated external beam radiotherapy (Experimental): Patients will receive 5 fractions of 7.25Gy per fraction which will be delivered alternate days over no more than 2 weeks to provide a total dose of 36.25Gy.
  Interventions: Radiation: Sterotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Brachytherapy — High Dose-Rate Brachytherapy
  Arms: High dose-rate brachytherapy
Radiation: Sterotactic Body Radiotherapy — Hypofractionated External Beam Radiotherapy
  Arms: Ultra-hypofractionated external beam radiotherapy

SUMMARY:
The RO-PIP trial aims to determine the feasibility of recruitment to a trial randomising patients to salvage ultra-hypofractionated external beam radiotherapy or high dose rate brachytherapy and provide prospective data on patient recorded toxicity outcomes that will inform a future phase III trial.

DETAILED DESCRIPTION:
Radiotherapy is the most common curative treatment for non-metastatic prostate cancer, however up to 13% of patients will develop local recurrence within 10 years. Patients can undergo further and potentially curative treatment including salvage surgery, brachytherapy (BT), external beam radiotherapy (EBRT), high intensity focused ultrasound and cryotherapy. Systematic review shows that high dose rate (HDR) BT and stereotactic body radiotherapy (SBRT) have the best outcomes in terms of biochemical control and lowest side effects. The RO-PIP trial aims to determine the feasibility of recruitment to a trial randomising patients to salvage HDR-BT or SBRT and provide prospective data on patient recorded toxicity outcomes that will inform a future phase III trial.

The primary endpoint of the RO-PIP feasibility study is to evaluate the patient recruitment potential over 2 years to a trial randomising to either SBRT or HDR-BT for patients who develop local recurrence of prostate cancer following previous radiation therapy. The aim is to recruit 60 patients across 3 sites over 2 years and randomise 1:1 to SBRT or HDR-BT. Secondary objectives include recording clinician and patient reported outcome measures (PROMs) to evaluate treatment-related toxicity. In addition, the study aims to identify potential imaging, genomic and proteomic biomarkers that are predictive of toxicity and outcome based on hypoxia status, a prognostic marker of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged over 18 years
* Histologically confirmed locally recurrent prostate cancer (following previous radiotherapy no less than 2 years ago)
* No metastatic disease
* Able and willing to provide an informed consent to participate
* World Health Organisation (WHO) performance status 0-2
* Reasonable urinary function (IPSS < 20 and Qmax > 10 ml/second on flow tests)
* Greater than 10 year life expectancy

Exclusion Criteria:

* Patients who are unfit for a general anaesthetic due to other comorbidities
* Clinical or radiological evidence of metastatic prostate disease
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent
* Contraindication or intolerance of magnetic resonance scanning
* Prior prostatectomy
* History of inflammatory bowel disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Treatment Feasibility | 24 months
  Recruitment rates for the whole 24-month recruitment period will be reported overall and per recruiting site. The average recruitment rate per month and in total over the formal monitoring period will be reported.

SECONDARY OUTCOMES:
Patient Reported Toxicity | 0-3 months and >3 months
  Incidence of patient reported acute (0-3 months) and long-term toxicity (>3 months) and impact on QoL determined by EPIC-26 (prostate cancer related QoL and functional outcomes), EORTC QLQ-C30 (general QoL score) and international prostate symptom score (IPSS) (urinary and sexual functional outcomes) measurements (Key secondary endpoint).
Clinician Reported Toxicity | 0-3 months and >3 months
  Incidence of clinician-reported treatment toxicity as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

OTHER OUTCOMES:
Imaging biomarkers | 1 month and 12 months
  MRI biomarkers at 1 month and 1 year post-treatment predictive of toxicity based on PROMs.
Imaging Reproducibility | Baseline, 1 and 12 months
  Multiple measures of image quality and reproducibility of prostate functional imaging (e.g. diffusion coefficient values from IVIM sequences) for measuring tumour biology will be summarised.
Hypoxia Gene Signature | Baseline
  Hypoxia levels based on a hypoxia associated gene signature obtained from the pre-salvage RT biopsy correlated with MRI biomarkers.
Proteomic Biomarkers | Baseline, 1, 3 and 6 months
  Changes in the levels of inflammatory cytokine signatures from urine and blood obtained at baseline and after reirradiation in relation to PROMs.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Henry, Principal Investigator — University of Leeds